CLINICAL TRIAL: NCT07121621
Title: PHArmaCokinetics of methYLphenidate in Adult Patients With Attention-Deficit /Hyperactivity Disorder: Comparison Between Patients With and Without OBesity
Brief Title: PHArmaCokinetics of methYLphenidate in Adult Patients With Attention-Deficit /Hyperactivity Disorder
Acronym: PHACYLOB
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DR240305; 2024-519461-22-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD); Obesity (Body Mass Index &Amp;Amp;gt;30 kg/m2); Methylphenidate; Obesity &Amp; Overweight
Keywords: Methylphenidate; Attention Deficit Hyperactivity Disorder (ADHD); Obesity; Pharmacokinetics
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Obesity; Overweight | interventions — Adiposity

STUDY DESIGN:
Intervention Model Description: The pharmacological intervention, which will be the same for all patients in the study, will consist in administering MPH at CIC 1415 (URHC of Tours) in the form of Prolonged Release at the patient's usual dosage, in the early morning.
  Compare the total area under the curve (AUC) of MPH and alpha-phenyl 2 piperidine acid (APP), its active metabolite, between patients with ADHD and obesity and patients with ADHD but without obesity.
  Pharmacokinetic study with repeated measurements at T0 (just before MPH administration) then T30 minutes, T1 hour, T2h, T3h, T4h, T6h, T8h (8 measurements) after MPH administration, in 15 patients with ADHD and obesity (BMI≥30 kg/m2) and in 15 patients with ADHD but without obesity (BMI<30 kg/m2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PHArmacoKinetics of methYLphenidate in adult patients with ADHD (Experimental): PHArmacoKinetics of methYLphenidate in adult patients with ADHD: patients with OBesity.
  PHArmacoKinetics of methYLphenidate in adult patients with ADHD: patients without OBesity.
  Interventions: Drug: PHArmacoKinetics of methYLphenidate in adult patients with ADHD: comparison between patients with and without OBesity.

INTERVENTIONS:
Drug: PHArmacoKinetics of methYLphenidate in adult patients with ADHD: comparison between patients with and without OBesity. — The pharmacological intervention, which will be the same for all patients in the study, will consist in administering MPH at CIC 1415 (URHC of Tours) in the form of Prolonged Release at the patient's usual dosage, in the early morning.
  Pharmacokinetic study with repeated measurements at T0 (just before MPH administration) then T30 minutes, T1 hour, T2h, T3h, T4h, T6h, T8h (8 measurements) after MPH administration, in 15 patients with ADHD and obesity (BMI≥30 kg/m2) and in 15 patients with ADHD but without obesity (BMI<30 kg/m2).

SUMMARY:
PHACYLOB PHArmaCokinetics of methYLphenidate in adult patients with Attention-Deficit Hyperactivity Disorder (ADHD) : comparison between patients with and without OBesity.

Its aim is to determine whether, for a comparable treatment dose, there are differences in the pharmacokinetic of methylphenidate between ADHD patients with obesitý and ADHD patients but without obesitý. More specifically, we will assess whether blood concentrations of methylphenidate (MPH; long acting form) are significantly higher or lower in either group at different times of the day.

To meet this objective, we are conducting this pharmacokinetic clinical trial with blood sampling and repeated clinical measurements just prior to MPH administration (= at T0) and then, at different times after administration, i.e. at times (T): T 30 minutes, T 1 hour, T2h, T3h, T4h, T6h, T8h after MPH administration. As far as MPH is concerned, this is the usual treatment. However, we may hypothesize that the distribution in the body may differ according to weight: hence the interest of this study

DETAILED DESCRIPTION:
The various phases of the study will take place at the Tours University Hospital:

* Patient selection (Department of Addictions): Eligibility assessment by the psychiatrist consulting patients with ADHD. Information regarding the study, risks, and constraints associated with the study.
* Patient inclusion (CIC 1415): Signed consent after informing the patient about the protocol, risks, and constraints. Collection of demographic and medical data, ADHD symptom intensity (ASRS-18), and individual psychological characteristics (emotional dysregulation: DERS-36, impulsivity: UPPS-P, binge eating disorder: BES).
* Clinical and laboratory assessments prior to MPH administration (CIC 1415): Blood pressure, NPF, serum creatinine, and complete liver function tests.
* MPH administration (CIC 1415): MPH LP is taken at the patient's usual dosage in the early morning.
* Repeated blood samples (CIC 1415) to measure plasma concentrations of MPH and APP before drug administration (T0), i.e., a pre-administration sample, then at T30 minutes (+/- 10 min), T1h (+/- 10 min), T2h (+/- 30 min), T3h (+/- 30 min), T4h (+/- 30 min), T6h (+/- 30 min), and T8h (+/- 30 min) after MPH administration. Clinical Research Nurses will accurately note the exact sampling times on the venous sampling accompanying sheets, including any differences from the theoretical schedule, in order to limit bias. Samples will be collected using sodium heparin trace element tubes, without separator gel (royal blue cap with black collar). These venous samples will be sent to and stored at the Biological Resources Center of Touraine (CRB-T). In addition, two aliquots must be taken and stored by the CRB-T. For each sample, one aliquot must be sent to the Medical Pharmacology Department and the second retained for safety.
* Assessment of perceived efficacy and tolerance of treatment (CIC 1415): visual analog scale allowing self-assessment of ADHD symptoms according to the patient at T0, T30 minutes, T1h, T2h, T3h, T4h, T6h, T8h and the effect on food craving; clinical assessment of treatment tolerance at T4h and T8h.
* Patient discharged home, in the absence of serious adverse side effects.
* Pharmacokinetic analysis and modeling (Medical Pharmacology Department): transfer from the CRB-T at the end of the study, plasma assays, pharmacokinetic modeling based on patient data.
* Note: For pharmacokinetic analysis, 6 mL of blood will be collected in sodium heparin tubes over the 8 sampling times. A total of 48 mL of blood will therefore be collected per patient on their day of participation. These samples will ultimately be destroyed after the results have been analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over
* Diagnosis of ADHD by a psychiatrist, based on DSM-5 criteria (ADHD mixed form, predominantly inattentive or predominantly hyperactive/impulsive)
* Treatment with methylphenidate LP (Ritaline) with a stable dosage for at least two weeks.
* BMI inclusion criteria: (1) for obese group: BMI ≥ 30 kg/m2; (2) for non-obese group: BMI < 30 kg/m2.
* Participant affiliated to a social security scheme
* Written consent signed by participant

Exclusion Criteria:

* Contraindications to methylphenidate treatment
* Treatment with an oral or nasal decongestant vasoconstrictor; association with a non-selective MAOI antidepressant.
* Treatment with a proton pump inhibitor within the last 2 weeks.
* Severe cognitive impairment (clinical evaluation)
* Severe alcohol use disorder, i.e. at least 6 DSM-5 criteria for substance use disorder (clinical evaluation)
* Known prior renal impairment
* Pregnant or breast-feeding women
* Female patients of childbearing age without at least one acceptable contraceptive method (see definition in Appendix 1)
* Patients under legal protection
* Inability of the patient to self-assess the intensity of ADHD symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-02 (Estimated); Study Completion 2026-09-02 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) of blood concentrations of MPH and APP, its active metabolite, measured up to 8 hours (T0, T30 minutes, T1h, T2h, T3h, T4h, T6h, T8h) after MPH administration, compared between patients with and without obesity. | Anticipated recruitment period: 12 months / Duration of each subject's participation: 1 day / Total duration of research: 12 months and 1 day
  The primary endpoint is the area under the curve (AUC) of blood concentrations of MPH and APP, its active metabolite, measured up to 8 hours (T0, T30 minutes, T1h, T2h, T3h, T4h, T6h, T8h) after MPH administration, compared between patients with and without obesity.

CONTACTS AND LOCATIONS:
Locations (1):
- Center Hospitalier Régional Universitaire of TOURS, Tours, Indre-et-Loire, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faraone SV, Banaschewski T, Coghill D, Zheng Y, Biederman J, Bellgrove MA, Newcorn JH, Gignac M, Al Saud NM, Manor I, Rohde LA, Yang L, Cortese S, Almagor D, Stein MA, Albatti TH, Aljoudi HF, Alqahtani MMJ, Asherson P, Atwoli L, Bolte S, Buitelaar JK, Crunelle CL, Daley D, Dalsgaard S, Dopfner M, Espinet S, Fitzgerald M, Franke B, Gerlach M, Haavik J, Hartman CA, Hartung CM, Hinshaw SP, Hoekstra PJ, Hollis C, Kollins SH, Sandra Kooij JJ, Kuntsi J, Larsson H, Li T, Liu J, Merzon E, Mattingly G, Mattos P, McCarthy S, Mikami AY, Molina BSG, Nigg JT, Purper-Ouakil D, Omigbodun OO, Polanczyk GV, Pollak Y, Poulton AS, Rajkumar RP, Reding A, Reif A, Rubia K, Rucklidge J, Romanos M, Ramos-Quiroga JA, Schellekens A, Scheres A, Schoeman R, Schweitzer JB, Shah H, Solanto MV, Sonuga-Barke E, Soutullo C, Steinhausen HC, Swanson JM, Thapar A, Tripp G, van de Glind G, van den Brink W, Van der Oord S, Venter A, Vitiello B, Walitza S, Wang Y. The World Federation of ADHD International Consensus Statement: 208 Evidence-based conclusions about the disorder. Neurosci Biobehav Rev. 2021 Sep;128:789-818. doi: 10.1016/j.neubiorev.2021.01.022. Epub 2021 Feb 4. PMID 33549739
- [Background] Brunault P, Frammery J, Montaudon P, De Luca A, Hankard R, Ducluzeau PH, Cortese S, Ballon N. Adulthood and childhood ADHD in patients consulting for obesity is associated with food addiction and binge eating, but not sleep apnea syndrome. Appetite. 2019 May 1;136:25-32. doi: 10.1016/j.appet.2019.01.013. Epub 2019 Jan 11. PMID 30641157